CLINICAL TRIAL: NCT02234011
Title: A Placebo-Controlled Crossover Trial of Intranasal Ketamine for the Treatment of Obsessive-Compulsive Disorder
Brief Title: A Trial of Intranasal Ketamine for the Treatment of Obsessive-Compulsive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to difficulty in recruiting participants.
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Brian P. Brennan, MD, M.D., Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2014P001140
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine/Placebo (Experimental): Participants in this group will receive 5 sprays (10 mg each) of intranasal ketamine for the first treatment visit, then receive 5 sprays of placebo (saline solution) at the second treatment visit two weeks later.
  Interventions: Drug: Ketamine; Drug: Placebo
- Placebo/Ketamine (Experimental): Participants in this group will receive 5 sprays of placebo (saline solution) for the first treatment visit, then receive 5 sprays (10 mg each) of intranasal ketamine at the second treatment visit two weeks later.
  Interventions: Drug: Ketamine; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine
Drug: Placebo

SUMMARY:
This study is being done to learn whether administration of intranasal (inhaled through the nose) ketamine reduces symptoms of obsessive-compulsive disorder (OCD). Ketamine has been approved by the U.S. Food and Drug Administration (FDA) as an anesthetic agent (a medicine to reduce pain during surgery and other procedures) but ketamine has not been approved by the FDA as a treatment for OCD.

The investigators believe that ketamine may be effective in reducing symptoms of OCD due to its ability to decrease the activity of a specific brain chemical called glutamate. Previous studies have shown that people with OCD can have abnormal levels of glutamate in their brains. This is the first time that intranasal ketamine is being studied in people with OCD. However, studies have been done in the past using intravenous (IV; through a needle into a vein in your arm) ketamine in people with OCD, and intranasal ketamine has been studied in people with other psychiatric conditions.

This research study will compare ketamine to placebo. The placebo looks exactly like ketamine, but contains no ketamine. At some time during the study, the investigators will give you ketamine. At another time, the investigators will give you placebo. Placebos are used in research studies to see if the results are due to the study drug or due to other reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥ 18 and ≤ 55
2. Meets DSM-IV50 criteria for OCD as the primary presenting diagnosis as determined by the investigator (participants with secondary comorbid dysthymia, major depression, anxiety disorders, eating disorders, and other obsessive-compulsive spectrum disorders will still be eligible for enrollment).
3. Score of ≥ 18 on the Y-BOCS at screening

Exclusion Criteria:

1. Unwillingness or inability to provide written informed consent.
2. Active suicidal ideation at screening
3. Lifetime history of psychotic disorder or autism spectrum disorder
4. DSM-IV diagnosis of alcohol or substance dependence, with the exception of nicotine dependence, within three months prior to screening
5. Any history of intolerance or hypersensitivity to ketamine
6. Any history of nasal/sinus anomalies or dysfunction (e.g., nasal obstruction or history of nasal surgery)
7. Clinically significant medical disease including, but not limited to, cardiac (including uncontrolled hypertension or uncontrolled hypotension, arrhythmias, congestive heart failure, angina), pulmonary, hepatic, renal, or endocrine disorders, which would increase the risk to the participant or interfere with interpretation of results as judged by the principal investigator.
8. Clinically significant neurologic disease including, but not limited to, seizure disorder, neurodegenerative diseases, transient ischemic attacks, neural vascular disease, stroke, cerebral aneurysms, and history of traumatic brain injury.
9. Female participants with a positive serum or urine pregnancy test at screening
10. Pregnancy. Females of childbearing potential must be using an effective contraceptive method (e.g., abstinence, prescription oral contraceptives, contraceptive injections, double-barrier method, male partner sterilization). Women that are not of childbearing potential are defined as: postmenopausal (>45 years of age with amenorrhea for at least 12 months, or any age with menorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level >40 IU/ml); permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy); or otherwise be incapable of pregnancy.
11. Female participants who are lactating.
12. Any screening laboratory abnormality deemed clinically significant by the investigator
13. Currently taking opiate pain medications, dextromethorphan, St. John's Wort, theophylline, or tramadol.
14. Any participation in an investigational drug trial within 30 days of enrollment in study.
15. Contraindication to having an MRI.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brennan, M.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject completed the screening visit, but chose to withdraw from study due to time commitment required. Because this subject only completed a screening visit, she was never entered into the treatment arm of the study (which begins at the baseline visit).
Groups:
- Treatment: No participants enrolled in treatment portion of study.
Period: Overall Study
Arm/Group | Treatment
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment: No participants enrolled in treatment portion of study, and therefore never completed a baseline visit. One subject completed a screening visit and then withdrew from study due to time commitments.
Arm/Group | Treatment
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Observing if Ketamine May Cause a Decrease in OCD Symptoms
Description: Examining if ketamine is associated with a decrease in OCD symptoms as measured by the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) at completion of one treatment when compared to placebo (saline solution).
  The Y-BOCS measures OCD symptoms on a scale of 0-40, with higher numbers indicating greater severity of OCD symptoms. For this study, subjects had to have a Y-BOCS of greater than or equal to 18 in order to participate.
Time Frame: Baseline to Week 5
Population: One subject had a screening visit, but was never enrolled in the treatment portion and therefore never had any sort of treatment analysis performed on her data.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Treatment: No participants enrolled in treatment portion of study. One subject had a screening visit, but since she never entered the treatment portion of the study and never received the study medication. Because she never had any exposure to the study medication and had no visits other than the initial screening visit, she was never at risk for any adverse events related to study medication.
  No adverse events related to study medication were collected since no subjects ever entered the treatment phase of this study.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No